CLINICAL TRIAL: NCT06075849
Title: A Multicenter, Open-label, Dose Escalation and Expansion, Phase I Study to Evaluate Safety, Tolerability, Pharmacokinetics, Pharmacodynamics, and Anti-tumor Activity of PB101 in Patients With Advanced Solid Tumor
Brief Title: Phase I Study to Evaluate Safety and Anti-tumor Activity of PB101, an Anti-angiogenic Immunomodulating Agent
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Panolos Bioscience (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PB101_101
Record Dates: First submitted 2023-09-25; First posted 2023-10-10 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Solid Tumor, Adult; Solid Tumor; Gastric Cancer; Hepatocellular Carcinoma; Metastatic Colorectal Cancer; Advanced Solid Tumor
Keywords: Neoplasms; Angiogenesis Inhibitors; Antineoplastic Agents; Angiogenesis Modulating Agents; Immuno Modulating Agents
MeSH Terms: conditions — Stomach Neoplasms; Carcinoma, Hepatocellular; Colorectal Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PB101 (Experimental): A total of 6 cohorts are planned, and each dose escalation will proceed in a traditional 3+3 scheme.
  Interventions: Drug: PB101

INTERVENTIONS:
Drug: PB101 — Cohorts of 3-6 patients receive PB101 until the MTD is determined. The dose (2 mg/kg-15 mg/kg) assigned to the cohort will be administered weekly for two 28-day cycles or until progressive disease (PD), unacceptable toxicity, withdrawal of subject consent, and/or the investigator's decision to discontinue the study treatment occurs.
  Administration may be continued for subjects in whom PB101 provides clinical benefits at the discretion of the investigator.

SUMMARY:
This clinical trial is designed as a multi-center, open-label, dose-escalation, dose-expansion, phase 1 clinical trial and will be evaluating the safety and efficacy of PB101 in patients with advanced solid tumors who have progressed after standard of care.

PB101 may stop the growth of tumor cells by blocking blood flow to the tumor and modulating the tumor microenvironment.

DETAILED DESCRIPTION:
Primary Objectives

To assess the safety and tolerability of PB101 and determine the maximum tolerated dose (MTD) and/or the recommended phase-2 dose

Secondary Objectives

1. To characterize the pharmacokinetics of PB101.
2. To identify the preliminary anti-tumor activity of PB101.
3. To assess the immunogenicity of PB101.

Tertiary Objectives

To explore the correlation between potential pharmacodynamic (PD) biomarkers (e.g., vascular endothelial growth factor(VEGF)-A, placental growth factor (PlGF) and VEGFR1 signaling) and anti-cancer activity of PB101.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following inclusion criteria.

1. ≥19 years of age
2. Patients with unresectable locally advanced or metastatic solid tumor, confirmed histologically and cytologically, who is refractory to existing standard of care or has progressive disease and has no other available standard of care available.
3. Patient who has at least one measurable or non-measurable but evaluable lesion that meets the RECIST version 1.1.
4. Patient whose expected survival period is 12 weeks or longer.
5. Patient with eastern cooperative oncology group (ECOG) performance status ≤ 2
6. Patient whose adequate hematological function, and kidney and liver functions have been confirmed by the following criteria. (Laboratory tests are allowed to re-conducted within the screening period.)
7. Patient with adequate anticoagulant functions according to the following criteria:

   * Without receiving anticoagulant therapy, patient whose international normalized ratio (INR) is ≤ 1.5 x upper limit of normal (ULN) and partial thromboplastin time (PTT) is ≤ 5 seconds above the ULN.
   * When receiving an oral anticoagulant or low molecular weight heparin, patient whose prothrombin time (PT) or PTT is confirmed to be stable for at least 2 weeks.
   * When receiving warfarin, patient whose INR is ≤3.0 There must be no active bleeding (bleeding within 14 days) or pathological conditions with a high risk of bleeding (e.g., tumor with macrovesicular invasion or known varicose vein).
8. Patient who voluntarily gave informed consent in writing to participate in this clinical trial after being provided with information on the nature and risks of the study as well as the expected desirable benefits and AEs of the investigative product (IP).

Exclusion Criteria:

Patients who meet any of the following criteria cannot participate in this clinical trial.

1. Patient expected to show hypersensitivity to the active ingredient and components of PB101 or similar drugs.
2. Patient with the following medical history (including surgery/procedure history) confirmed.

   * Major surgery within 4 weeks prior to administration of the IP, and clinically significant traumatism.
   * Cardiovascular disease (including unstable angina, myocardial infarction, stroke, and transient ischemic attack), congestive heart failure (NYHA class III or IV), or clinically significant arrhythmia uncontrollable by medication within 24 weeks prior to administration of the IP.
   * Patient whose left ventricular ejection fraction (LVEF) measured by echocardiography, multigated blood pool scan (MUGA) scan or the standard procedure at the institution before administration of the IP is less than the lower limit of normal at the institution. However, if there is no reference LVEF set at the institution, 50% will be treated as the reference level.
   * Vascular disorders (e.g., deep vein thrombosis, pulmonary embolism, aortic aneurysm, and peripheral arterial thrombosis) within 24 weeks prior to administration of the IP
   * Life-threatening (Grade 4) venous thromboembolism (regardless of the duration, even if it is a past medical history)
   * Medical history of primary malignancies other than indication for this clinical trial. However, the following cases are allowed:

     * Not less than 3 years have passed since the cure diagnosis of a primary malignancy. However, in case of papillary thyroid cancer, patients who underwent curative resection can participate in the study regardless of the duration.
     * At least 1 year has passed since complete resection of cutaneous basal cell carcinoma/squamous cell carcinoma of the skin or successful treatment of cervical carcinoma in situ.
   * Psychiatric disorder that may significantly affect the participation in the study at the discretion of the investigator.
3. Patient with the following comorbidities confirmed at the time of participation in the study.

   * Squamous cell carcinoma of the lung (current and past medical history).
   * Interstitial lung disease or pulmonary fibrosis (current and past medical history).
   * The following hemorrhage-related and digestive system diseases (current and past medical history).

     * Evidence of active bleeding, hemorrhagic diathesis, coagulopathy, and tumor with macrovesicular invasion.
     * Clinically significant medical history of digestive system, such as peptic ulcer, gastrointestinal bleeding, gastrointestinal or non-gastrointestinal fistulas or perforations, intra-abdominal abscesses, clinical symptoms and signs of gastrointestinal obstruction, and inflammatory bowel disease.
   * Clinically significant pericardial effusion, pleural fluid, or ascites. However, in case of ascites, patients who do not require paracentesis for improvement of the symptoms can participate in the study.
   * Uncontrolled hypertension (systolic blood pressure (SBP) > 150 or diastolic blood pressure (DBP) > 90 mmHg even after medication).
   * Infection of active hepatitis B* or C† virus

     *Hepatitis B surface antigen (HBsAg)-positive at screening. However, for HBsAg positive, not excluded if the patient is taking antiviral agents stably.

     †Hepatitis C virus antibody (HCV Ab)-positive at screening. However, if the result of HCV RNA test is negative, participation is possible.
   * Human immunodeficiency virus (HIV)-positive.
   * Severe infection or other uncontrolled active infection that requires administration of systemic antibiotics, antivirals, etc. at the discretion of the investigator
   * New or active brain metastases. However, patients who do not need central nervous system (CNS) treatment immediately (or within 1 cycle) at the discretion of the investigator can participate in the study.
   * Leptomeningeal metastasis
   * Serious and unhealed wound or fracture
4. Patient who received the following treatment regimens (drug/non-drug)

   * patient who received the following anti-cancer treatments other than this IP.

     * Chemotherapy, hormone therapy, and radiation therapy within 2 weeks prior to administration of the IP. However, patients who completed local radiotherapy as a palliative therapy for the purpose of pain relief in areas other than the target lesion (e.g., site of bone metastases) and recovered from following acute toxicity (e.g., myelosuppression).However, patients who completed local radiotherapy as a palliative therapy for the purpose of pain relief in areas other than the target lesion (e.g., site of bone metastases) and recovered from following acute toxicity (e.g., myelosuppression).However, patients who completed local radiotherapy as a palliative therapy for the purpose of pain relief in areas other than the target lesion (e.g., site of bone metastases) and recovered from following acute toxicity (e.g., myelosuppression).
     * Targeted therapies or immunotherapy within 4 weeks prior to administration of the IP.
     * Administration history of nitrosoureas or mitomycin-C within 6 weeks prior to administration of the IP.
   * Administration history of nonsteroidal anti-inflammatory drugs (NSAID) and anti-platelet agents within 7 days prior to administration of the IP. However, for aspirin, doses of 325 mg/day are allowed.
5. Patient who participated in another clinical study within 4 weeks prior to administration of the IP and received (underwent procedure of) an investigational drug (or medical device).
6. Patient who continues to experience a clinically significant toxicity or adverse event of Grade 2 or higher (based on NCI-CTCAE v5.0) after prior anti-cancer therapy. However, hair loss (any grade) and neuropathy (Grade 2 or lower) are exceptions.
7. Pregnancy test positive at screening, or pregnant or lactating woman.
8. Female or male subject of childbearing potential who does not agree to stay abstinent or use an effective method of contraception† during the study period and for at least 26 weeks (women) or 14 weeks (men) after the last dose of the IP.

   †Effective method of contraception:
   * Hormonal contraceptive: Subdermal implants, injections, oral contraceptives, etc. However, in case of ovarian/breast cancer, hormonal contraception is not allowed.
   * Implantation of an intrauterine device or intrauterine system: Loop, and hormone-containing intrauterine system.
   * Sterilization procedure or surgery of the subject or his/her spouse (partner): Vasectomy, tubal ligation, etc.
9. Other patients deemed ineligible to participate in the study by the investigator.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-10-25 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | 8 weeks
  Frequency by dose group
Permanent discontinuation / dose reduction due to adverse events (AE) | 8 weeks
  Frequency and percentage by dose group due to adverse drug reactions (ADR)
Adverse events | 8 weeks
  Incidence by dose group for treatment-emergent adverse events (TEAEs), ADRs, serious adverse events (SAEs), and serious ADRs
Electrocardiogram (ECG) | 8 weeks
  Clinically significant changes in ECG results compared to baseline
Left ventricular ejection fraction (LVEF) | 8 weeks
  Multigated blood pool scan (MUGA) or echocardiography (ECHO), clinical significance and significant changes evaluated

SECONDARY OUTCOMES:
Objective response rate (ORR) | 8 weeks
  Frequency according to response evaluation criteria in solid tumors (RECIST) v1.1
Duration of response (DOR) | 8 weeks
  Time analyzed using Kaplan-Meier method
Progression free survival (PFS) | 8 weeks
  Time analyzed using Kaplan-Meier method
Disease control rate (DCR) | 8 weeks
  Time analyzed using Kaplan-Meier method
Time to progression (TTP) | 8 weeks
  Time analyzed using Kaplan-Meier method
Overall survival (OS) | 8 weeks
  Time analyzed using Kaplan-Meier method
Tumor Evaluations | 8 weeks
  Tumor response will be evaluated according to RECIST v1.1

OTHER OUTCOMES:
Area under the concentration-time curve (AUC) | 8 weeks
  AUC last, AUC inf
Maximum plasma concentration (Cmax) | 8 weeks
  For each time point by dose group, number of subjects, mean, standard deviation, and median, minimum, and maximum values will be presented for continuous variables, and frequency and percentage will be presented for categorical variables.
Minimum plasma concentration (Cmin) | 8 weeks
  For each time point by dose group, number of subjects, mean, standard deviation, and median, minimum, and maximum values will be presented for continuous variables, and frequency and percentage will be presented for categorical variables.
Time to Cmax (Tmax) | 8 weeks
  For each time point by dose group, number of subjects, mean, standard deviation, and median, minimum, and maximum values will be presented for continuous variables, and frequency and percentage will be presented for categorical variables.
Terminal half-life (t1/2) | 8 weeks
  For each time point by dose group, number of subjects, mean, standard deviation, and median, minimum, and maximum values will be presented for continuous variables, and frequency and percentage will be presented for categorical variables.
Biomarkers | 8 weeks
  Serum vascular endothelial growth factor (VEGF) - A, placental growth factor (PlGF), and VEGF receptor 1 (VEGFR1) measurements by dose group and visit
Immunogenicity | 8 weeks
  Anti-PB101 antibody analysis

CONTACTS AND LOCATIONS:
Overall Officials: Hong Jae Chon, MD/PhD, Principal Investigator — CHA University Bundang Medical Center; Keun Wook Lee, MD/PhD, Principal Investigator — Seoul National University Bundang Hospital; Myung-Ah Lee, MD/PhD, Principal Investigator — The Catholic University of Korea
Locations (3):
- South Korea (3):
  - CHA University Bundang Medical Center, Seongnam
  - Seoul National University Bundang Hospital, Seongnam
  - The Catholic University of Korea Seoul St. Mary's Hospital, Seoul

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee JE, Kim C, Yang H, Park I, Oh N, Hua S, Jeong H, An HJ, Kim SC, Lee GM, Koh GY, Kim HM. Novel glycosylated VEGF decoy receptor fusion protein, VEGF-Grab, efficiently suppresses tumor angiogenesis and progression. Mol Cancer Ther. 2015 Feb;14(2):470-9. doi: 10.1158/1535-7163.MCT-14-0968-T. Epub 2014 Dec 22. PMID 25534360
- [Background] Go EJ, Yang H, Lee SJ, Yang HG, Shin JA, Lee WS, Lim HS, Chon HJ, Kim C. PB101, a VEGF- and PlGF-targeting decoy protein, enhances antitumor immunity and suppresses tumor progression and metastasis. Oncoimmunology. 2023 Sep 20;12(1):2259212. doi: 10.1080/2162402X.2023.2259212. eCollection 2023. PMID 37744990
- See also: Company link — https://www.panolos.com
- See also: Mechanism of Action — https://www.youtube.com/watch?v=HPGW7sunrsI